CLINICAL TRIAL: NCT01477073
Title: A Phase I, Mono-center, Placebo and Comparator Controlled, Single-blind, Randomized, Parallel Group, Clinical Study to Determine Multiple Dose Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of FSH-GEX(TM) Administered Subcutaneously in Healthy Pituitary-suppressed Female Volunteers
Brief Title: Multiple Dose FSH-GEX(TM) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Collaborators: Glycotope Biotechnology GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEXGP24102
Record Dates: First submitted 2011-11-09; First posted 2011-11-22 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Female Infertility
Keywords: in-vitro fertilization; reproductive disorder
MeSH Terms: conditions — Infertility, Female | interventions — follitropin alfa; Urofollitropin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- FSH-GEX 75 IU (Experimental): follitropin epsilon 75 IU QD
  Interventions: Drug: FSH-GEX™
- FSH-GEX 150 IU (Experimental): follitropin epsilon 150 IU QD
  Interventions: Drug: FSH-GEX™
- FSH-GEX 150 IU QAD (Experimental): follitropin epsilon 150 IU QAD
  Interventions: Drug: FSH-GEX™
- recombinant FSH (Active Comparator): Gonal-f 150 IU QD
  Interventions: Drug: recombinant FSH
- urinary FSH (Active Comparator): Bravelle 150 IU QD
  Interventions: Drug: urinary FSH
- Placebo (Placebo Comparator): Placebo QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FSH-GEX™
  Other Names: follitropin epsilon
  Arms: FSH-GEX 150 IU; FSH-GEX 150 IU QAD; FSH-GEX 75 IU
Drug: recombinant FSH
  Other Names: Gonal-f
  Arms: recombinant FSH
Drug: urinary FSH
  Other Names: Bravelle
  Arms: urinary FSH
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of the current study is the pharmacokinetic and pharmacodynamic characterization of a multiple dose administration of FSH-GEX™ in healthy pituitary-suppressed female volunteers, in comparison with two marketed comparator products or placebo.

DETAILED DESCRIPTION:
Healthy pituitary-suppressed female subjects received multiple doses of FSH-GEX at one of 2 different dose levels (75 IU and 150 IU dosing once daily (QD), or 150 IU (dosing once every other day (QAD)) for maximal 7 Days. They were compared with subjects who received a urinary FSH or a recombinant FSH or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects from 18-40 years of age at screening.
2. Subjects must be in good health as determined by medical and gynecological history, physical and gynecological examination, vital signs, body measurements, electrocardiogram, and laboratory tests
3. Subjects must be willing to use additional non-hormonal contraception
4. Subjects must have used a combined oral contraceptive, combined contraceptive vaginal ring or combined contraceptive patch
5. Vital signs which are within the following ranges: systolic blood pressure between 90-140 mmHg, diastolic blood pressure between 50-90 mmHg, pulse rate between 40 - 100 bpm
6. Subjects must have a body weight of minimally 50.0 kg with a BMI between 18.0 and 29.9 kg/m2
7. Able to provide written informed consent prior to study participation.
8. Able to communicate well with the investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Smokers of more than 5 cigarettes per day.
2. Average daily intake of more than 3 units of alcohol per day (where 1 unit equals 250 mL of beer, 125 mL of wine or 25 mL of spirits) or an average weekly intake of more than 21 units alcohol.
3. Use of any prescription drug or over-the-counter medication from screening until the end-of-study visit, without prior approval of the investigator. Paracetamol® is acceptable without prior approval.
4. Any drugs that may reduce the effectiveness of combination oral contraceptive (COC) from screening until the end-of-study visit
5. Administration of any investigational product or use of any investigational device within 30 days prior to Screening.
6. Donation or loss of 500 mL or more of blood within 90 days prior to first dosing of FSH-GEX(TM).
7. History of acute or chronic bronchospastic disease
8. History of allergies for drugs, seafood, nuts, eggs, wasp-stings; history of atopic allergy. A known hypersensitivity to any of the study drugs.
9. Any surgical or medical condition which might alter the absorption, distribution, metabolism, or excretion of drugs or which may jeopardize the subject in case of participation in the study.
10. History or presence of any malignancy.
11. Determined or suspected pregnancy.
12. Breast feeding women.
13. History of (or current) endocrine abnormalities
14. Contraindication for the use of oral contraceptives
15. Contraindication for the use of follitropin alfa, follicle-stimulating hormone (FSH) or any of the excipients (hypersensitivity to follitropin alfa, FSH or any of the excipients; tumors of the hypothalamus or the pituitary gland; ovarian enlargement or cyst not due to polycystic ovarian disease; gynecological bleeding of unknown origin; ovarian, uterine, or mammary carcinoma).
16. Porphyria or family history of porphyria.
17. History of ovarian surgery.
18. Any ovarian or abdominal abnormality that would interfere with adequate ultrasound investigation.
19. An abnormal cervical smear
20. History or presence of an immune-compromising disease, or a positive human immunodeficiency virus (HIV) test result in the past or at the screening visit.
21. History of Hepatitis B or C, or a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at the screening visit.
22. History of drug or alcohol abuse within the 12 months prior to the screening visit or evidence of such abuse
23. Planned surgery or hospitalization during the period of the study.
24. Concurrent participation or participation within 30 days before screening in another clinical trial, or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study or previous participation in the 104676-CS0160 (FSH-GEXTM) study.
25. Injection of one or more doses of any depot contraceptive drug /drug combination ≤10 months prior to screening.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of FSH-GEX™ following multiple dose administration by subcutaneous injection | 43 days
  frequency of dose related adverse events, measurement of vital signs, body measurements, transvaginal ultrasound, ECG and laboratory values in comparison to placebo and the two comparators with marketing authorization

SECONDARY OUTCOMES:
pharmacokinetic profile of FSH-GEX™ following multiple dose administration by subcutaneous injection (part 1) | 28 time points up to 14 days post-dose
  Peak Plasma Concentration (Cmax)
pharmacokinetic profile of FSH-GEX™ following multiple dose administration by subcutaneous injection (part 2) | 28 time points up to 14 days post-dose
  Area under the plasma concentration versus time curve (AUC)
pharmacodynamic parameters of FSH-GEX™ following multiple dose administration by subcutaneous injection | 17 time points up to 14 days post-dose
  Estradiol (E2), Luteinizing Hormone (LH) and inhibin B serum levels
pharmacodynamic parameters of FSH-GEX™ following multiple dose administration by subcutaneous injection | 9 time points up to14 days post-dose
  follicular response and endometrial thickness as determined by transvaginal ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Glycotope GmbH Director, Study Director — Glycotope GmbH
Locations (1):
- Glycotope Investigational Site, Groningen, Netherlands

REFERENCES:
- [Result] Abd-Elaziz K, Duijkers I, Stockl L, Dietrich B, Klipping C, Eckert K, Goletz S. A new fully human recombinant FSH (follitropin epsilon): two phase I randomized placebo and comparator-controlled pharmacokinetic and pharmacodynamic trials. Hum Reprod. 2017 Aug 1;32(8):1639-1647. doi: 10.1093/humrep/dex220. PMID 28591833